CLINICAL TRIAL: NCT05574595
Title: The Effect of Self-selected Soothing Music on Fistula Puncture-related Pain and Comfort in Hemodialysis Patients
Brief Title: Effect on Pain and Comfort Associated With Fistula Puncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Aylin Aydin Sayilan, Associate Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022/4
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Hemodialysis Patients
Keywords: pain; comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Mean of the Hemodialysis Comfort Scale scores of the experimental and group patients (Experimental): To the Experimental Group; The information form and the short form of the comfort scale will be applied to the patient who is taken to the dialysis unit to start HD treatment.
  Interventions: Other: Music theraphy
- The mean of the Hemodialysis Comfort Scale scores of the control group patients (No Intervention): No procedure was performed on the patients in the control group.

INTERVENTIONS:
Other: Music theraphy — In each session, the desired type of music will be played approximately 6 minutes before the procedure (Shabandokht-Zarmi et al., 2017). After the end of the music, the cannulation process will be performed by the dialysis nurse. The level of pain experienced by the patient immediately after needle insertion into the fistula will be evaluated with VAS by a research-independent nurse working in the dialysis unit.
  Other Names: There is no other name.
  Arms: The Mean of the Hemodialysis Comfort Scale scores of the experimental and group patients

SUMMARY:
Purpose This study was carried out as the design of the targeted design in terms of targeting and comfort in the patient with hemodialysis.

Material and Methods: It was successfully tested both in the control team of a hospital at the point of sale in Turkey and with experience. By block randomization method to randomize. Data were collected with "Patient identification formula", "Visual Analog Scale (VAS)" and "Hemodialysis Comfort Scale". Independent sample t-test was used in the analysis of the data, analysis of variance in repeated measurements and Cohen'd was used to calculate the size.

DETAILED DESCRIPTION:
It is appropriate to suggest a non-pharmacological rather clinical rather than a literature-free method, al. Also, due to the fact that the duration of anesthetic effect will expire from the dialysis treatment used (Subramanian et al., 2012).

Participant's care continues for inappropriate pain management. This quality standard is one of the criteria of a standard rather than a preference for a simple, reliable and inexpensive non-pharmacological choice.

As far as investigators know, there are very few studies investigating the effect of a patient's choice of music on pain following insertion of a needle into a fistula in hemodialysis patients. More focused on non-pharmacological types such as pharmacological and aromatherapy. Therefore, the aim of this study was to examine the effect of the type of music chosen by hemodialysis patients on pain and comfort associated with fistula puncture.

ELIGIBILITY:
Inclusion Criteria:

* be volunteering,
* 18 years or older,
* receiving hemodialysis treatment for at least 6 months
* not any hearing problem.

Exclusion Criteria:

* have hearing problem
* not be volunteering.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
The Efficacy of Music on Pain Level | 7 days
  Visual Analog Scale

SECONDARY OUTCOMES:
The Efficacy of Music on Comfort Level | 7 days
  Comfort Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nurşen KULAKAÇ, pHD, Principal Investigator — Gümüşhane Universıty

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayilan S, Sayilan AA, Kulakac N. The effect of self-selected soothing music on fistula puncture-related pain and comfort levels in hemodialysis patients: a randomized controlled, single-blind, single-center study. Int Urol Nephrol. 2025 Oct 28. doi: 10.1007/s11255-025-04877-5. Online ahead of print. PMID 41148531